CLINICAL TRIAL: NCT01004900
Title: Comparison of Selective Laser Trabeculoplasty With Prostaglandin Analogues for Lowering Intraocular Pressure in Eyes With Primary Angle Closure Glaucoma
Brief Title: Intraocular Pressure (IOP) Lowering Effect of Selective Laser Trabeculoplasty Versus Prostaglandin Analogues in Angle Closure Glaucoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: A/ Prof Aung Tin, A/ PROF & CONSULTANT, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R657/07/2009
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Glaucoma
Keywords: Glaucoma, Angle Closure; Selective laser trabeculoplasty; Primary Angle Closure Disease
MeSH Terms: conditions — Glaucoma; Glaucoma, Angle-Closure | interventions — Travoprost; Timolol; brinzolamide; Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabeculoplasty (Active Comparator)
  Interventions: Procedure: Selective Laser Trabeculoplasty
- Control (Medication) (Active Comparator)
  Interventions: Drug: Travoprost/ Timolol/ Azopt/ Brimonidine

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty — This is a laser procedure used to treat glaucoma by reducing the pressure in the eye. SLT works by using laser light to stimulate the body's own healing response to lower your eye pressure. Using a special wavelength and energy, the laser affects only pigmented (melanin containing) cells of your eye. SLT improves the flow of fluid in the eye, which in turn lowers your eye pressure.
  Arms: Trabeculoplasty
Drug: Travoprost/ Timolol/ Azopt/ Brimonidine — Travoprost (Topical eye drops) administered once daily before sleep
  Arms: Control (Medication)

SUMMARY:
Glaucoma affects 66 million people worldwide and is the leading cause of irreversible blindness, and Primary angle-closure glaucoma (PACG) is a major form of glaucoma in Asia.

Laser peripheral iridotomy (LPI) has been advocated as the first line treatment in all cases of PACG. In addition to relieving the relative pupil block element of the condition, it can open up the drainage angle, alleviating appositional and synechial angle-closure and in the long-term this may control intraocular pressure (IOP) and prevent progression of glaucomatous optic neuropathy. However recent data indicate that iridotomy is not successful in controlling IOP in the long term, and the majority of cases develop a clinically significant rise in IOP requiring medical therapy or surgery.

Laser trabeculoplasty has been a recognized treatment option for Primary open angle glaucoma (POAG) since the 1980s. Recently a more selective and less destructive method of performing laser trabeculoplasty has evolved. Selective Laser Trabeculoplasty (SLT) specifically targets the pigmented trabecular meshwork cells without producing collateral damage and destruction to adjacent structures. Morphologic study performed on human autopsy eyes treated with SLT noted no structural or collateral thermal damage to the trabecular beams in the uveal and corneoscleral meshwork. As SLT specifically has its effect on the targeted pigmented trabecular meshwork it is unlikely to generate PAS. It may be a useful treatment option for PACG patients in whom the angle has widened following laser peripheral iridotomy.

The proposed study is a randomized controlled trial to assess the effectiveness of SLT in reducing IOP in cases of PACG in which the angle has opened up following LPI, but IOP remains high(>21 mmHg). 100 subjects will be randomized to receive either SLT or medical treatment to achieve IOP control. They will be followed up for 6 months.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND PURPOSE

The aim of this study is to determine whether selective laser trabeculoplasty (SLT) is an effective treatment for lowering intraocular pressure (IOP) in patients with primary angle closure glaucoma (PACG), compared to prostaglandin analogues, the current first choice IOP-lowering medical therapy.

STUDY DESIGN The study design for this project is a prospective randomized controlled trial. It will not be possible to blind either the subject or observer to the intervention due to the use of laser in the intervention group and medical therapy in the control group. Subjects will then be followed-up for 6 months

STUDY POPULATION

The study population will be patients with primary angle closure glaucoma attending the Singapore National Eye Centre, who fulfil the inclusion criteria and are willing to take part in the study.

WASH OUT REGIMEN: for patients already on medication

Eligible patients who are already on one or two-glaucoma medications are required to complete a washout period before being randomized. Washout periods will vary according to the previous medication used and are as follows:

Prostaglandin analogues 4 weeks Beta blockers 3 weeks Adrenergic agonist 2 weeks Cholinergic agonist 5 days Carbonic Anhydrase Inhibitors 5 days

Pre-study washout period check Patients who are on prostaglandin analogues or beta blockers prior to the study will be required to undergo a washout period of 3 and 4 weeks respectively prior to the study. For this group of patients, there will be a safety check during the second week. Patients whose IOP>30 mm hg during this washout check will be stopped from further washout and be withdrawn from the study.

Treatment of subjects

PLANNED INTERVENTION

Selective laser trabeculoplasty procedure The laser procedure will be performed on all patients as follows

* A drop of Brimonidine will be instilled into the eye to be treated 15 minutes prior to the procedure.
* Topical anaesthesia will be administered and the Latina SLT lens and coupling fluid will be used for the procedure.
* The slit-lamp attached to the laser will be focused on the full height of the trabecular meshwork.
* The laser power will be set to 0.6mJ and increased in 0.1mJ steps until small champagne -like bubbles appear from the treated area of the trabecular meshwork. The laser spot size would be 400µm.
* Approximately 60-120 non-overlapping shots will be placed onto at least 180 degrees of the trabecular meshwork that is visible and without PAS. More non-overlapping shots can be placed if sufficient extent of the trabeculum is visible.

Post - laser the patient will be given a one week course of topical Prednisolone forte four times a day for the treated eye.

Intraocular pressure will be checked 30-60 minutes after the procedure. IOP spikes of ≥ 5mmHg or to a level of ≥ 28mmHg will be treated with Diamox if not contraindicated.

Intraocular pressure will be checked one week post SLT. If the IOP ≥28mmHg, tablet diamox will be given for 3 days.

Retreatment of SLT If IOP remains elevated, one further treatment of SLT will be given to the patient. This treatment will be administered either at the four week or three month follow up visit.

If there is a <20% reduction of IOP from baseline either at the week 4 or month 3 follow-up visit, then SLT will be repeated using the same laser parameters as described above. The patient will be seen again one week after the repeated laser treatment.

IIf the IOP is <21mmHg or there is >20% reduction of IOP from baseline at at the week 4 or month 3 follow-up visit, then no further treatment will be given to the patient.

IOP will be checked one week after repeat SLT. If the IOP is still high (>24 mmHg), treatment modification will be provided (see Treatment Modification below).

Control group Those patients randomized to the control group will be commenced on topical treatment to lower the IOP. The agent for lowering IOP will be a prostaglandin analogue, Travoprost, which will be applied once a day at night.

A stepwise addition of Timolol 0.5%, dorzolamide or brimonidine will be implemented until IOP is controlled (see below Treatment Modification).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary angle closure or primary angle closure glaucoma with documented pre-LPI angle closure of ≥180 degrees of the angle (Trabecular meshwork not visible in primary position using gonioscopy)
* One month post LPI, angle has opened up (visibility of trabecular meshwork) for at least 180 degrees of the angle
* Intraocular pressure between 21-≤30 mmHg without treatment following LPI OR Intraocular pressure between 21-≤30 mmHg after wash out regimen as described below for patients who are already medications following LPI.
* Informed Consent
* Age more than 21 years

Exclusion Criteria:

* Secondary causes of angle closure like subluxed lens, uveitis, trauma and neovascular glaucoma
* Presence of advanced sight-threatening glaucoma defined as vertical cup-disc ratio > 0.9 or visual field constriction involving <100 of the central visual field performed with the Humphrey Visual Field Analyzer II using the SITA STD algorithm with a 24-2 test pattern.
* Cataract that is deemed significant enough to require surgery during the course of the trial or that makes field testing or optic disc imaging not technically possible- visual acuity less than 20/40 due to any type of cataract.
* Previous intraocular surgery, SLT, ALT, refractive surgery or iridoplasty.
* Documented previous history of angle closure.
* Use of contact lens
* Chronic use of topical or systemic steroids
* Participation in another therapeutic drug study within the last 30 days
* Severe health problems precluding follow-up such as end-stage heart disease, kidney disease, respiratory disease, or cancer and life expectancy less than one year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | 6 months
  Fluid pressure inside the eye

CONTACTS AND LOCATIONS:
Overall Officials: Tin Aung, FRCOphth, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Derived] Narayanaswamy A, Leung CK, Istiantoro DV, Perera SA, Ho CL, Nongpiur ME, Baskaran M, Htoon HM, Wong TT, Goh D, Su DH, Belkin M, Aung T. Efficacy of selective laser trabeculoplasty in primary angle-closure glaucoma: a randomized clinical trial. JAMA Ophthalmol. 2015 Feb;133(2):206-12. doi: 10.1001/jamaophthalmol.2014.4893. PMID 25429421